CLINICAL TRIAL: NCT05254587
Title: Accuracy of IOLMASTER 700 Total Keratometry (TK) in Patients Undergoing Post-Laser Vision Correction Cataract Surgery
Brief Title: Accuracy of IOLMASTER 700 Total Keratometry (TK)
Status: Completed | Type: Observational
Sponsor: Advanced Vision Care (Other)
Collaborators: Clinical Research Consultants, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AVC-005
Record Dates: First submitted 2022-02-15; First posted 2022-02-24 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Myopia; Hyperopia; Cataract
Keywords: Laser Vision Correction; Cataract Surgery
MeSH Terms: conditions — Myopia; Hyperopia; Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Retrospective
  Interventions: Device: IOLMASTER 700 TK
- Prospective
  Interventions: Device: IOLMASTER 700 TK

INTERVENTIONS:
Device: IOLMASTER 700 TK — 4 different intraocular lens (IOL) calculation methods (Haigis TK, ASCRS calculator, Barrett True K Classic K, Barrett True K TK) will be performed using the preoperative biometry and post operative refraction data.

SUMMARY:
This is a multicenter study to compare the accuracy of IOL calculations in post-laser vision corrected eyes that are about to undergo or have undergone cataract surgery.

DETAILED DESCRIPTION:
This is a multicenter study to compare the accuracy of IOL calculations using 4 different IOL calculation methods (Haigis TK, ASCRS calculator, Barrett True K with classic K, and Barrett True K TK) performed using the preoperative biometry data from post-laser vision correct eyes that are about to undergo or have undergone cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, 18 years of age or older at the time of cataract surgery.
2. Patient has had LVC and IOL cataract surgery within 3 years or is scheduled to undergo IOL cataract surgery performed for the treatment of visually significant cataracts.

   Note: The only IOLs permitted for use in this study are Monofocal (ZCBOO, LI61AO, SN60WF, SA60WF, MX60E) and Toric Lenses (Tecnis 2 ZCU, ZCT, SN6ATx, SA6ATx, MX60ET).
3. Best corrected distance visual acuity (BCDVA) potential of 20/30 or better (as measured by Retinal Acuity Meter (RAM) or Potential Acuity Meter (PAM).
4. Patients who have a manifest refraction that is myopic or hyperopic after previous LVC.
5. Patients that have biometric measurements (including Axial Length) for the IOL cataract surgery that were performed preoperatively with the IOLMaster700, including Barrett True K /TK.
6. Signed and received a copy of the signed written informed consent (pertain to the prospective subjects only).
7. For prospective patients, willingness and ability to comply with schedule for follow-up visits and postoperative evaluations.

Exclusion Criteria:

1. Patients with a history of any of the following:

   1. Corneal pathology - Epithelial Basement Membrane Dystrophy (EMBD), Irregular Astigmatism, Decentered LASIK/PRK, Radial Keratotomy (RK), Fuchs Dystrophy
   2. Retinal pathology - Visually significant Epiretinal Membrane (ERM) with loss of foveal contour, Large/ Medium Drusen, Cystoid Macular Edema (CME), History of Retinal Detachment
   3. Optic neuropathy
   4. Advanced glaucoma
   5. Amblyopia
   6. Strabismus
   7. Relative Afferent Pupillary Defect (RAPD) indicating an optic neuropathy.
2. Patients with a previous history of small incision lenticule extraction (SMILE) surgery and/or glaucoma filtering procedure (defined as tubes or trabeculectomy) other than photorefractive keratectomy (PRK) or LASIK.
3. Patient who had to undergo A-scan measurement to retrieve Axial Length (AL) values.
4. Patient has had LVC and IOL cataract surgery within 3 years or is scheduled to undergo IOL cataract surgery performed for the treatment of visually significant cataracts with the presence or intention of implanting a multifocal, extended depth of focus, accommodating and light adjustable lens (such as, but not limited to, TFAT / TFNT; DAT / DFT; ICB00/DIB/DIU/DAT; ZXT; DFW; SN6AD1; AT-50; RxSIGHT).
5. Patients in whom the study eye experiences any intraoperative surgical complications or complex cataract surgeries (vitrectomy, corneal suturing).
6. Patients with previous LVC where one eye was treated for myopia and the other eye was treated for hyperopia.
7. Patient is participating in another study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Subjects that have had laser vision correction and cataract surgery (retrospective cohort) or have had laser vision correction surgery and are scheduled for cataract surgery (prospective cohort).
Sampling Method: Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2024-01-27 (Actual); Study Completion 2024-01-27 (Actual)

PRIMARY OUTCOMES:
Total Keratometry Accuracy Assessment | 4 Weeks
  Subjects utilizing Total Keratometry within (+/- 0.50 D, +/- 0.75 D, +/- 1.00 D) compared to the proportion of subjects utilizing traditional keratometry readings.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Fram, MD, Principal Investigator — Advanced Vision Care
Locations (7):
- United States (7):
  - Empire Eye & Laser Center, Bakersfield, California
  - Advanced Vision Care, Los Angeles, California
  - Wolstan & Goldberg Eye Associates, Torrance, California
  - Solomon Eye Physicians and Surgeons, Bowie, Maryland
  - Ophthalmic Partners PC, Bala-Cynwyd, Pennsylvania
  - MUSC Storm Eye Institute29425, Charleston, South Carolina
  - Virginia eye consultant, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No